CLINICAL TRIAL: NCT01088295
Title: Metabolic Abnormalities, Telmisartan and HIV Infection
Brief Title: HIV and Fat Accumulation
Acronym: MATH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: California HIV/AIDS Research Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MATH
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: HIV Infection
Keywords: Metabolic; HIV; Fat accumulation; AIDS; Metabolic abnormalities in HIV infection; HIV Infections
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telmisartan (Experimental): Telmisartan 40mg po daily for 24 weeks
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan
  Other Names: Micardis

SUMMARY:
This is a research study to see whether fat accumulation either under the skin or in the body's organs, for example, the liver, improves in men and women who take a drug called telmisartan. The investigators will be looking at how the amount of fat in the body changes when HIV-positive persons on effective anti-HIV therapy take telmisartan. The investigators will be using a CT scan to make this comparison. Telmisartan is not an HIV medication. It is a medication used to treat blood pressure, but has been shown to decrease fat in the organs in people both with and without high blood pressure. The study involves 8 visits over a period of about 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive men and women 18 years and older
* HIV-1 infection as documented by ELISA and confirmed by Western blot or plasma HIV-1 RNA >2000 on two occasions
* Documented central fat accumulation
* HIV RNA documented to be less than 50 copies/mL at screening and undetectable by assay of choice for at least 12 weeks prior to entry
* Current antiretroviral therapy with a suppressive, highly active antiretroviral regimen.
* Systolic BP >115mmHg.
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Pregnancy (current or within the last 6 months) or nursing
* Uncontrolled hypertension
* Prohibited concomitant medications
* Subjects with untreated hyperlipidemia must be willing to abstain from initiating therapy for the 24 week duration fo the study.
* Subjects undergoing treatment for diabetes with oral hypoglycemic agents must be willing to remain on their current dose of insulin sensitizing agents for the duration of the study.
* Known, untreated renal artery stenosis
* Unstable coronary artery disease/angina or decompensated congestive heart failure.
* Any history of intolerance to any member of the angiotensin receptor blocker class of agents.
* Need for ongoing potassium supplementation.
* Screening laboratory values as follows ANC (absolute neutrophil count) <750 cells/mm3 Hemoglobin <10 gm/dL ClCr (creatinine clearance)< 30 ml/min (estimated by Cockcroft-Gault equation) AST (aspartate aminotransferase) or ALT (alanine aminotransferase) > 3 x ULN (upper limit of normal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Lake, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA CARE Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Lake JE, Tseng CH, Currier JS. A pilot study of telmisartan for visceral adiposity in HIV infection: the metabolic abnormalities, telmisartan, and HIV infection (MATH) trial. PLoS One. 2013;8(3):e58135. doi: 10.1371/journal.pone.0058135. Epub 2013 Mar 14. PMID 23516440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between May and October 2010 at the UCLA CARE Center.
Period: Overall Study
Arm/Group | Telmisartan
Started | 36
Completed | 35
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Telmisartan
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Median Change in Visceral Adipose Tissue (VAT) Volume
Description: VAT volume was quantified at each timepoint by L4-L5 single slice computed tomography
Time Frame: Baseline and 24 weeks
Population: as-treated analysis
Measure: Median (Inter-Quartile Range); unit: cm^2
Arm/Group | Telmisartan
Number analyzed (Participants) | 35
cm^2 | -4.6 [-29.5 to 31.2]

ADVERSE EVENTS:
Arm/Group | Telmisartan
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No